CLINICAL TRIAL: NCT05301764
Title: An Open Label, Phase Ib/II Trial of LVGN6051 Combined with Anlotinib in the Treatment of Locally Advanced, Metastatic or Recurrent Refractory Soft Tissue Sarcoma
Brief Title: A Study of LVGN6051 Combined with Anlotinib in Patient with Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lyvgen Biopharma Holdings Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVGN6051-301
Record Dates: First submitted 2022-03-02; First posted 2022-03-31 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LVGN6051 combined with Anlotinib (Experimental): LVGN6051 Dose Escalation in the combination treatment with Anlotinib
  Interventions: Combination Product: LVGN6051 and Anlotinib

INTERVENTIONS:
Combination Product: LVGN6051 and Anlotinib — LVGN6051: Route of administration is IV infusion, and the frequency of administration is once every 3 weeks(Q3W). One cycle is 3 weeks, and treatment can be up to 35 cycles if patients receive benefits. Anlotinib: Rout of administration is oral. The initial dose of anlotinib was 12 mg for subjects with body surface area ≥ 1.5m2 and 10 mg for subjects with body surface area < 1.5m2. If the subjects in the combined treatment group were not tolerated, the dose of anlotinib was reduced to 10 mg for subjects with body surface area ≥ 1.5m2 and 8 mg for subjects with body surface area < 1.5m2.
  One cycle is 3 weeks, including oral for 2 weeks and withdrawal for 1 week.

SUMMARY:
The purpose of this study is to asess the safety and tolerability and efficacy of LVGN6051 combined with anlotinib in patient with soft tissue sarcoma.

DETAILED DESCRIPTION:
This is a phase 1b/II, open-label, multicenter study of LVGN6051 combined with anlotinib in patients with locally advanced, metastatic or recurrent refractory soft tissue sarcoma.

The study is comprised of a dose escalation phase (Ib) to determine the RP2D and an expansion phase (II) to further explore the safety and efficacy of combination treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years, who was histologically or cytologically diagnosed unresectable locally advanced, metastatic or recurrent refractory soft tissue sarcoma.
2. Ability to understand and willingness to sign a written informed consent document (ICF). Informed consent of subjects must be performed before the study, and the written informed consent shall be voluntarily signed by himself or his guardian; The subject or his guardian can communicate well with the investigator, and perform according to the protocol.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
4. Estimated life expectancy, in the judgment of the Investigator, of at least 90 days.
5. Adequate bone marrow function, as defined by all of the following:

   1. hemoglobin (Hb) ≥ 90 g/L, and
   2. absolute neutrophil count (ANC) ≥ 1.5x109/L, and
   3. platelet count (PLT) ≥ 75x109/L.
6. Adequate liver function, as defined by all of the following:

   1. Total bilirubin ≤ 1.5 × ULN; or ≤ 2.5 × ULN for patients who have serum bilirubin increases due to underlying Gilbert's Syndrome or familial benign unconjugated hyperbilirubinemia.
   2. Aspartate Aminotransferase (AST) ≤ 1.5 × ULN, and Alanine Transaminase (ALT) ≤ 1.5× ULN.
   3. International normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤ 1.5×ULN, for subjects who are receiving anticoagulant therapy, INR level should be within therapeutic range.
   4. Amylase and lipase ≤1.5 × ULN
7. Adequate renal function as defined by an estimated serum creatinine clearance of ≥ 50 mL/min (calculated by Cockcroft-Gault formula) or serum creatinine≤1.5×ULN.
8. Women of childbearing potential must agree to abstain from heterosexual intercourse or use highly effective contraceptive methods from the time of signing informed consent and through 120 days after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she (or her partner) is participating in this study, she should inform her research physician immediately.

   a. A woman of childbearing potential is any woman, regardless of sexual orientation, who meets the following criteria: 1. has not undergone tubal ligation, a hysterectomy, or bilateral oophorectomy; or 2. has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
9. Men enrolled on this study must agree to abstain, be surgically sterilized, or agree to use highly effective methods of contraception, including barrier contraception from the time of signing informed consent and through 120 days after the last dose of study drug.
10. Patients should recover from all reversible clinically significant AEs of previous anticancer therapies to baseline or NCI-CTCAE v. 5.0 Grade 0-1, except for alopecia (any Grade), Grade < 2 sensory or motor peripheral neuropathy, lymphopenia, or hypothyroidism on hormone replacement (Grade 2), within 14 days prior to the first dose on study. Inclusion of patients with other toxicities deemed not clinically significant (Grade ≤ 2) should be discussed and approved by the Medical Head of Sponsor.
11. All patients must have at least one measurable lesion as defined by RECIST v1.1 for solid tumors.
12. All patients with advanced/metastatic soft tissue sarcoma receiving LVGN6051 combinated with Anlotinib must have received one prior line of approved chemotherapy and disease progresses or intolerance confirmed by imaging examination before enrollment. Approved chemotherapy must include anthracycline, except acinar soft tissue sarcoma and clear cell sarcoma, which can be included in patients with recurrence or metastasis who are newly diagnosed or who only receive surgical treatment.

Exclusion Criteria:

1. Prior therapy with anti-CD137 therapy.
2. Receipt of systemic anticancer therapy including investigational agents or devices within 5 half-lives of the first dose of study treatment. For anticancer therapies with half-life greater than 5 days, a washout of 28 days or longer is acceptable
3. The subject was experienced radiotherapy within 14 days before the first dose of study treatment. [Previous radiotherapy to the central nervous system (CNS) within 28 days of the first dose of study treatment].
4. Known unstable CNS metastasis and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically and radiographically stable, without evidence of recurrence/progression, have no evidence of new or enlarging brain metastases or cephaledema, and are using no corticosteroids for at least 7 days prior to study medication.
5. Received a live-virus vaccine within 30 days of the first dose of study drug.
6. Grade ≥ 3 allergic reaction to treatment with a monoclonal antibody or has a known or suspected hypersensitivity to components of the study treatment(s).
7. Baseline QT interval corrected by Fridericia's formula (QTcF) > 480 milliseconds or known to have congenital prolonged QT syndrome.
8. History of Grade ≥ 3 immune-related AEs (irAEs). Exceptions: hypothyroidism, type 1 diabetes mellitus (Type 1 DM), and dermatologic irAEs (patients with previous Steven Johnson Syndrome, toxic epidermal necrolysis or other severe forms of dermatitis are ineligible) are allowed. Type 1 DM should be controlled with HbA1c <8% as per ADA recommendation.
9. Receiving an immunologically based treatment for any reason, including chronic use of systemic steroids equivalent to > 10 mg/day of prednisone within 7 days of the first dose of study drug or at any time during study participation.

   Note: Use of inhaled or topical steroids or systemic corticosteroids equivalent to ≤ 10 mg/day prednisone equivalent is permitted as is short-term use of corticosteroids at doses equivalent to > 10 mg/day of prednisone (e.g., pre-medication prior to contrast).
10. Treatment with systemic immune-stimulatory agents (e.g., IL-2, IFNγ) within 4 weeks prior to the first dose of study drug.
11. History or current active or chronic autoimmune disease including but not limited to inflammatory bowel disease, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis that has required systemic treatment in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease.

    Exception: Patients with vitiligo or resolved childhood asthma/atopy, hypothyroidism on stable hormone replacement, controlled asthma, Type I diabetes, Graves' disease, Hashimoto's disease, or with Medical Monitor approval.
12. Clinically significant cardiac condition, including unstable angina, acute myocardial infarction within 6 months of Cycle 1 Day 1, New York Heart Association Class III or IV congestive heart failure, unstable angina pectoris or arrhythmia requiring therapy.

    Note: A patient with an arrhythmia may enroll if the patient is on antiarrhythmic medication and is in a rate- controlled rhythm on the screening electrocardiogram (ECG).
13. Pleural effusion or pericardial effusion with uncontrolled or requiring repeat drainage (recurrence within two weeks after intervention), or recurrent ascites requiring drainage ≥ once a month.
14. Active infection requiring intravenous (IV) anti-infectives within 14 days before the first dose of study treatment, or nonhealing wound or ulcer.
15. Current evidence or history of interstitial lung disease or active, noninfectious pneumonitis requiring treatment such as oral or intravenous glucocorticoids.
16. Female patients who are pregnant or breastfeeding (confirmation that the patient is not pregnant must be by a negative serum pregnancy test result obtained during screening; pregnancy testing is required of women of childbearing potential but not required for postmenopausal or surgically sterilized women).
17. Any evidence of severe or uncontrolled systemic disease including, but not limited to, active bleeding diathesis, organ transplantation.
18. Subjects with known positive test results of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
19. Subjects with known active hepatitis B [hepatitis B surface antigen (HBsAg) positive] and / or hepatitis B core antibody (HBcAb) positive and hepatitis B virus DNA (HBV DNA) ≥ 104 copies/ml or 2000IU/ml) or hepatitis C virus RNA (HCV RNA) positive were known
20. Any other disease or clinically significant abnormality in laboratory parameters, including serious medical or psychiatric illnesses/conditions, which in the judgment of the Investigator might compromise the safety of the patient, integrity of the study, interfere with the patient participation in the study, or compromise the study objectives.
21. Previously received an allogeneic tissue/organ transplant, stem cell or bone marrow transplant or solid organ transplant.
22. Previous cell therapy (including but not limited to Car T cell therapy).
23. The investigator believes subject has other acute or serious or chronic medical or psychological diseases and he is not suitable to participate in the clinical trial.
24. Traditional Chinese medicine containing anticancer ingredients or with clear anticancer indications has been used in the past (auxiliary drugs were not included), and the elution period is 30 days.
25. Other malignant tumors ≤5 years before the first dose. Exceptions are: early stage malignancies that have been radically cured (carcinoma in situ or stage I tumours), such as carcinoma in situ of the cervix, basal cell or squamous cell skin cancers that have been adequately treated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-03-19 (Estimated); Study Completion 2025-10-19 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of LVGN6051 combined with Anlotinib and to recommend the Phase II dose | Up to 24 months
  To evaluate the safety and tolerability of LVGN6051 combined with Anlotinib through evaluation of the frequency and severity of AEs, serious adverse events(SAEs)
To characterize the safety and tolerability of LVGN6051 combined with Anlotinib and to recommend the Phase II dose | At the end of Cycle 1 (each cycle is 21 days)
  To evaluate the safety and tolerability of LVGN6051 combined with Anlotinib through evaluation of the type of dose-limiting toxicities (DLTs)
to determine objective response rate (ORR) of phase II | Up to 24 months
  To assess the preliminary efficacy of LVGN6051 combined with Anlotinib in terms of objective response rate (ORR).

SECONDARY OUTCOMES:
To characterize the safety and tolerability of LVGN6051 combined with Anlotinib | Up to 24 months
  To evaluate the safety and tolerability of LVGN6051 combined with Anlotinib through evaluation of the frequency and severity of AEs, Treatment-emergent Adverse Events (TEAEs), immune-related AEs (irAEs), treatment-related adverse events TRAEs), and laboratory results, Vital Signs, Physical examinations.
To assess preliminary efficacy on overall survival (OS)(for Phase II only) using LVGN6051 combined with Anlotinib | Up to 24 months
  To assess the preliminary efficacy of LVGN6051 combined with Anlotinib in terms of overall survival (OS)(for Phase II only)
To assess preliminary efficacy on progression-free survival (PFS) using LVGN6051 combined with Anlotinib | Up to 24 months
  To assess the preliminary efficacy of LVGN6051 combined with Anlotinib in terms of progression-free survival (PFS)
To assess preliminary efficacy on duration of response (DoR) using LVGN6051 combined with Anlotinib | Up to 24 months
  To assess the preliminary efficacy of LVGN6051 combined with Anlotinib in terms of duration of response (DoR)
To assess preliminary efficacy on disease control rate (DCR) using LVGN6051 combined with Anlotinib | Up to 24 months
  To assess the preliminary efficacy of LVGN6051 combined with Anlotinib in terms of disease control rate (DCR)
To assess whether the anti-drug antibody (ADA) of LVGN6051 exist or not | Up to 24 months
  To evaluate the ADA of LVGN6051 by the number of ADA cases and incidence of ADA.
To characterize the PK (Pharmacokinetic) profile of LVGN6051 | Up to 24 months
  PK exposure parameters derived from plasma concentrations of LVGN6051
To explore the biomarkers based on the tumor tissue sample | Up to 24 months
  To explore the correlation between biomarkers and antitumor efficacy, including PD-L1 (programmed cell death-Ligand 1), MSI/dMMR (Microsatellite Instability/Deficient Mismatch Repair), TMB (Tumor Mutation Burden).
To explore the biomarker IL-6 (interleukin- 6) based on the serum samples. | Up to 15 days
  To explore the changes of biomarker IL-6 (interleukin- 6) after LVGN6051 and anlotinib treatment
To explore the biomarker IL-12 (interleukin- 12) based on the serum samples. | Up to 15 days
  To explore the changes of biomarker IL-12 (interleukin- 12) after LVGN6051 and anlotinib treatment
To explore the biomarker TNF-α (Tumor Necrosis Factor-α) based on the serum samples. | Up to 15 days
  To explore the changes of biomarker TNF-α (Tumor Necrosis Factor-α) after LVGN6051 and anlotinib treatment
To explore the biomarker IFN-γ (Interferon Gamma) based on the serum samples. | Up to 15 days
  To explore the changes of biomarker IFN-γ (Interferon Gamma) after LVGN6051 and anlotinib treatment
To explore the biomarker CD137 (also known as 4-1BB) based on the serum samples. | Up to 15 days
  To explore the changes of biomarker CD137 (also known as 4-1BB) after LVGN6051 and anlotinib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Hu, Principal Investigator — Shanghai 6th People's Hospital
Locations (5):
- China (5):
  - Henan cancer hospital, Zhenzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No